CLINICAL TRIAL: NCT01971424
Title: Assessment of Physical Performance After Oral Supplementation of Magnesium in a Sample of Old Women in Good Health
Acronym: Magnesium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Giuseppe Sergi, Medical Doctor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2011491
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Age Related Muscle Loss
Keywords: magnesium; SPPB; strength; physical performance; 24 hour magnesuria
MeSH Terms: interventions — Magnesium Oxide; Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mg oxide (Experimental): Participants were supplemented for 12-weeks with 300 mg of daily oral magnesium oxide.
  Interventions: Dietary Supplement: Mg oxide; Other: healthy diet
- Controls (No Intervention): The control group was educated by a trained dietician to follow a healthy diet.

INTERVENTIONS:
Dietary Supplement: Mg oxide
  Other Names: Magnesium oxide
  Arms: Mg oxide
Other: healthy diet
  Arms: Mg oxide

SUMMARY:
Magnesium deficiency is associated also in the elderly with low physical performance; nevertheless trials about the effect of supplementation of magnesium on physical performance are not available in old people. The aim of our study is to investigate whether 12-weeks of oral magnesium supplementation improves physical performance in healthy elderly women

ELIGIBILITY:
Inclusion Criteria:

* People over 65 years, not residents in nursing home, in good health

Exclusion Criteria:

* previous supplementation of calcium, potassium or magnesium
* use of pump proton inhibitors or digitalis
* important co-mordidities such renal failure

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes in short physical performance battery (SPPB) | Baseline and after 12 weeks

SECONDARY OUTCOMES:
Changes in appendicular skeletal mass (ASMMI) | Baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Geriatrics Division, Department of Medicine, Padua, Padova, Italy

REFERENCES:
- [Background] Dominguez LJ, Barbagallo M, Lauretani F, Bandinelli S, Bos A, Corsi AM, Simonsick EM, Ferrucci L. Magnesium and muscle performance in older persons: the InCHIANTI study. Am J Clin Nutr. 2006 Aug;84(2):419-26. doi: 10.1093/ajcn/84.1.419. PMID 16895893
- [Derived] Veronese N, Berton L, Carraro S, Bolzetta F, De Rui M, Perissinotto E, Toffanello ED, Bano G, Pizzato S, Miotto F, Coin A, Manzato E, Sergi G. Effect of oral magnesium supplementation on physical performance in healthy elderly women involved in a weekly exercise program: a randomized controlled trial. Am J Clin Nutr. 2014 Sep;100(3):974-81. doi: 10.3945/ajcn.113.080168. Epub 2014 Jul 9. PMID 25008857